CLINICAL TRIAL: NCT00406536
Title: Phase II Study: LYM-X-SORB™, an Organized Lipid Matrix: Fatty Acids and Choline in CF
Brief Title: Study of LYM-X-SORB™ to Improve Fatty Acid and Choline Status in Children With CF and PI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanti Polar Lipids, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Walter A. Shaw, Ph.D, Principle Investigator, Avanti Polar Lipids, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DK60302; R44DK060302 (NIH); 2R44DK060302-02A1 (NIH)
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Pancreatic Insufficiency; LYM-X-SORB™; LXS
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Lym-X-Sorb powder
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Lym-X-Sorb powder — Lym-X-Sorb is an organized matrix of lyso phosphatidylcholine (LPC), free fatty acid (FFA) and monoglyceride formulated at 20wt% with flour and sugar. A dosage contains 32 grams of powder and is consumed with food twice a day (6 to 11.9 years old) or three times per day (12 to 17.9 years old) for 18 months.
  Arms: 1
Dietary Supplement: Placebo powder — The placebo is composed of soybean oil, sunflower oil, fully hydrogenated cottonseed oil and flax seed oil dispersed at 16wt% on flour and sugar. The placebo is >99% triglycerides with no trans fatty acids. The fatty acid composition and caloric content is designed to match the active supplement (Lym-X-Sorb). A dosage contains 32 grams of powder and is consumed with food twice a day (6 to 11.9 years old) or three times per day (12 to 17.9 years old) for 18 months.
  Arms: 2

SUMMARY:
The purpose of this phase II research study is to evaluate the effectiveness of the next generation LYM-X-SORB™ in improving the essential fatty acid (EFA) and choline status for children and adolescents with Cystic Fibrosis (CF) and pancreatic insufficiency (PI).

DETAILED DESCRIPTION:
Fat malabsorption is common in individuals with cystic fibrosis (CF) and pancreatic insufficiency (PI). This places them at risk for caloric, essential fatty acid, and choline deficiency, which may in turn, lead to growth failure and a poorer clinical course. The purpose of this research study is to find whether or not taking LYM-X-SORB™ over an 18-month period, every day, will correct the problem people with CF and PI have with absorbing fat and choline. Participation will help CF doctors and other healthcare professionals learn more about the potential benefits of LYM-X-SORB™ to children and adolescents with CF and PI. These benefits may include better absorption of fat, better choline status, better growth in height, weight, muscle and bone, better lungs, and improvement of health status.

The study will enroll a total of 78 participants from Children's Hospital of Philadelphia (CHOP) and from several other Cystic Fibrosis Centers. One half of the participants will be randomly picked to receive the active powder with the LYM-X-SORB™ supplement and one half will receive a placebo (with no active supplement).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having cystic fibrosis (CF) with pancreatic insufficiency (PI)
* Subjects aged 6 to 17 years of age
* In usual state of good health
* Family and subject commitment to the 18-month study protocol
* Fecal elastase < 15µg/g stool

Exclusion Criteria:

* Forced expiratory volume at one second, % predicted (FEV1) < 40% predicted
* Other chronic health conditions that may affect GI absorption, growth, dietary intake, nutritional status
* Liver disease, lung transplant, celiac disease, allergy/intolerance to wheat/gluten, pregnant
* Participation in another CF nutrition-related intervention study
* Regular intake of fatty acids (i.e., fish oils) or choline nutritional supplements
* Home parenteral lipid administration (i.e., intralipids)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Improvements in essential fatty acid (EFA) and choline status over a 12-month period. | 12-month period

SECONDARY OUTCOMES:
Improvements in growth, nutritional, and pulmonary status over an 18-month period. | 18-month period

CONTACTS AND LOCATIONS:
Overall Officials: Walter A. Shaw, PhD, Principal Investigator — Avanti Polar Lipids, Inc.; Virginia A. Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Freedman SD, Blanco PG, Zaman MM, Shea JC, Ollero M, Hopper IK, Weed DA, Gelrud A, Regan MM, Laposata M, Alvarez JG, O'Sullivan BP. Association of cystic fibrosis with abnormalities in fatty acid metabolism. N Engl J Med. 2004 Feb 5;350(6):560-9. doi: 10.1056/NEJMoa021218. PMID 14762183
- [Background] Innis SM, Davidson AG, Chen A, Dyer R, Melnyk S, James SJ. Increased plasma homocysteine and S-adenosylhomocysteine and decreased methionine is associated with altered phosphatidylcholine and phosphatidylethanolamine in cystic fibrosis. J Pediatr. 2003 Sep;143(3):351-6. doi: 10.1067/S0022-3476(03)00326-3. PMID 14517519
- [Background] Chen A, Innis S. Assessment of phospholipid malabsorption by quantification of fecal phospholipid. J Pediatr Gastroenterol Nutr. 2004 Jul;39(1):85-91. doi: 10.1097/00005176-200407000-00017. PMID 15187787
- [Background] Chen AH, Innis SM, Davidson AG, James SJ. Phosphatidylcholine and lysophosphatidylcholine excretion is increased in children with cystic fibrosis and is associated with plasma homocysteine, S-adenosylhomocysteine, and S-adenosylmethionine. Am J Clin Nutr. 2005 Mar;81(3):686-91. doi: 10.1093/ajcn/81.3.686. PMID 15755840
- [Background] Lepage G, Yesair DW, Ronco N, Champagne J, Bureau N, Chemtob S, Berube D, Roy CC. Effect of an organized lipid matrix on lipid absorption and clinical outcomes in patients with cystic fibrosis. J Pediatr. 2002 Aug;141(2):178-85. doi: 10.1067/mpd.2002.124305. PMID 12183711
- [Background] Roulet M, Frascarolo P, Rappaz I, Pilet M. Essential fatty acid deficiency in well nourished young cystic fibrosis patients. Eur J Pediatr. 1997 Dec;156(12):952-6. doi: 10.1007/s004310050750. PMID 9453380
- [Background] Kalivianakis M, Verkade HJ. The mechanisms of fat malabsorption in cystic fibrosis patients. Nutrition. 1999 Feb;15(2):167-9. doi: 10.1016/s0899-9007(98)00155-5. No abstract available. PMID 9990588
- [Background] KUO PT, HUANG NN, BASSETT DR. The fatty acid composition of the serum chylomicrons and adipose tissue of children with cystic fibrosis of the pancreas. J Pediatr. 1962 Mar;60:394-403. doi: 10.1016/s0022-3476(62)80065-1. No abstract available. PMID 14460644
- [Background] Farrell PM, Mischler EH, Engle MJ, Brown DJ, Lau SM. Fatty acid abnormalities in cystic fibrosis. Pediatr Res. 1985 Jan;19(1):104-9. doi: 10.1203/00006450-198501000-00028. PMID 3918287
- [Background] Lloyd-Still JD, Johnson SB, Holman RT. Essential fatty acid status and fluidity of plasma phospholipids in cystic fibrosis infants. Am J Clin Nutr. 1991 Dec;54(6):1029-35. doi: 10.1093/ajcn/54.6.1029. PMID 1957818
- [Background] van Egmond AW, Kosorok MR, Koscik R, Laxova A, Farrell PM. Effect of linoleic acid intake on growth of infants with cystic fibrosis. Am J Clin Nutr. 1996 May;63(5):746-52. doi: 10.1093/ajcn/63.5.746. PMID 8615359
- [Background] Lepage G, Paradis K, Lacaille F, Senechal L, Ronco N, Champagne J, Lenaerts C, Roy CC, Rasquin-Weber A. Ursodeoxycholic acid improves the hepatic metabolism of essential fatty acids and retinol in children with cystic fibrosis. J Pediatr. 1997 Jan;130(1):52-8. doi: 10.1016/s0022-3476(97)70310-x. PMID 9003851
- [Background] Lloyd-Still JD, Bibus DM, Powers CA, Johnson SB, Holman RT. Essential fatty acid deficiency and predisposition to lung disease in cystic fibrosis. Acta Paediatr. 1996 Dec;85(12):1426-32. doi: 10.1111/j.1651-2227.1996.tb13947.x. PMID 9001653
- [Background] Strandvik B, Gronowitz E, Enlund F, Martinsson T, Wahlstrom J. Essential fatty acid deficiency in relation to genotype in patients with cystic fibrosis. J Pediatr. 2001 Nov;139(5):650-5. doi: 10.1067/mpd.2001.118890. PMID 11713441
- [Background] Gibson RA, Teubner JK, Haines K, Cooper DM, Davidson GP. Relationships between pulmonary function and plasma fatty acid levels in cystic fibrosis patients. J Pediatr Gastroenterol Nutr. 1986 May-Jun;5(3):408-15. doi: 10.1097/00005176-198605000-00013. PMID 3723260
- [Background] Biggemann B, Laryea MD, Schuster A, Griese M, Reinhardt D, Bremer HJ. Status of plasma and erythrocyte fatty acids and vitamin A and E in young children with cystic fibrosis. Scand J Gastroenterol Suppl. 1988;143:135-41. doi: 10.3109/00365528809090234. PMID 3164500
- [Background] Congden PJ, Bruce G, Rothburn MM, Clarke PC, Littlewood JM, Kelleher J, Losowsky MS. Vitamin status in treated patients with cystic fibrosis. Arch Dis Child. 1981 Sep;56(9):708-14. doi: 10.1136/adc.56.9.708. PMID 7294874
- [Background] Farrell PM, Bieri JG, Fratantoni JF, Wood RE, di Sant'Agnese PA. The occurrence and effects of human vitamin E deficiency. A study in patients with cystic fibrosis. J Clin Invest. 1977 Jul;60(1):233-41. doi: 10.1172/JCI108760. PMID 874086
- [Background] Freedman SD, Katz MH, Parker EM, Laposata M, Urman MY, Alvarez JG. A membrane lipid imbalance plays a role in the phenotypic expression of cystic fibrosis in cftr(-/-) mice. Proc Natl Acad Sci U S A. 1999 Nov 23;96(24):13995-4000. doi: 10.1073/pnas.96.24.13995. PMID 10570187
- [Background] Steinkamp G, Demmelmair H, Ruhl-Bagheri I, von der Hardt H, Koletzko B. Energy supplements rich in linoleic acid improve body weight and essential fatty acid status of cystic fibrosis patients. J Pediatr Gastroenterol Nutr. 2000 Oct;31(4):418-23. doi: 10.1097/00005176-200010000-00016. PMID 11045840
- [Background] Henderson WR Jr, Astley SJ, McCready MM, Kushmerick P, Casey S, Becker JW, Ramsey BW. Oral absorption of omega-3 fatty acids in patients with cystic fibrosis who have pancreatic insufficiency and in healthy control subjects. J Pediatr. 1994 Mar;124(3):400-8. doi: 10.1016/s0022-3476(94)70362-0. PMID 8120709
- [Background] McKeon-O'Malley C, Siwek D, Lamoureux JA, Williams CL, Kowall NW. Prenatal choline deficiency decreases the cross-sectional area of cholinergic neurons in the medial septal nucleus. Brain Res. 2003 Jul 11;977(2):278-83. doi: 10.1016/s0006-8993(03)02599-x. PMID 12834888
- [Background] Brandner C. Perinatal choline treatment modifies the effects of a visuo-spatial attractive cue upon spatial memory in naive adult rats. Brain Res. 2002 Feb 22;928(1-2):85-95. doi: 10.1016/s0006-8993(01)03363-7. PMID 11844475
- [Background] Yen CL, Mar MH, Craciunescu CN, Edwards LJ, Zeisel SH. Deficiency in methionine, tryptophan, isoleucine, or choline induces apoptosis in cultured cells. J Nutr. 2002 Jul;132(7):1840-7. doi: 10.1093/jn/132.7.1840. PMID 12097657
- [Background] James SJ, Miller BJ, Basnakian AG, Pogribny IP, Pogribna M, Muskhelishvili L. Apoptosis and proliferation under conditions of deoxynucleotide pool imbalance in liver of folate/methyl deficient rats. Carcinogenesis. 1997 Feb;18(2):287-93. doi: 10.1093/carcin/18.2.287. PMID 9054620
- [Background] da Costa KA, Cochary EF, Blusztajn JK, Garner SC, Zeisel SH. Accumulation of 1,2-sn-diradylglycerol with increased membrane-associated protein kinase C may be the mechanism for spontaneous hepatocarcinogenesis in choline-deficient rats. J Biol Chem. 1993 Jan 25;268(3):2100-5. PMID 8420980
- [Background] HANDLER P, BERNHEIM F. Choline deficiency in the hamster. Proc Soc Exp Biol Med. 1949 Dec;72(3):569-71. doi: 10.3181/00379727-72-17502. No abstract available. PMID 15400800
- [Background] Buchman AL, Dubin MD, Moukarzel AA, Jenden DJ, Roch M, Rice KM, Gornbein J, Ament ME. Choline deficiency: a cause of hepatic steatosis during parenteral nutrition that can be reversed with intravenous choline supplementation. Hepatology. 1995 Nov;22(5):1399-403. PMID 7590654
- [Background] Mason JB. Biomarkers of nutrient exposure and status in one-carbon (methyl) metabolism. J Nutr. 2003 Mar;133 Suppl 3(3):941S-947S. doi: 10.1093/jn/133.3.941S. PMID 12612180
- [Background] Roy CC, Weber AM, Morin CL, Lepage G, Brisson G, Yousef I, Lasalle R. Hepatobiliary disease in cystic fibrosis: a survey of current issues and concepts. J Pediatr Gastroenterol Nutr. 1982;1(4):469-78. doi: 10.1097/00005176-198212000-00005. PMID 7186061
- [Background] Weizman Z, Durie PR, Kopelman HR, Vesely SM, Forstner GG. Bile acid secretion in cystic fibrosis: evidence for a defect unrelated to fat malabsorption. Gut. 1986 Sep;27(9):1043-8. doi: 10.1136/gut.27.9.1043. PMID 3758817
- [Background] Roy CC, Weber AM, Morin CL, Combes JC, Nussle D, Megevand A, Lasalle R. Abnormal biliary lipid composition in cystic fibrosis. Effect of pancreatic enzymes. N Engl J Med. 1977 Dec 15;297(24):1301-5. doi: 10.1056/NEJM197712152972401. PMID 917086
- [Background] Weber AM, Roy CC, Morin CL, Lasalle R. Malabsorption of bile acids in children with cystic fibrosis. N Engl J Med. 1973 Nov 8;289(19):1001-5. doi: 10.1056/NEJM197311082891903. No abstract available. PMID 4742200
- [Background] Ulane MM, Butler JD, Peri A, Miele L, Ulane RE, Hubbard VS. Cystic fibrosis and phosphatidylcholine biosynthesis. Clin Chim Acta. 1994 Oct 31;230(2):109-16. doi: 10.1016/0009-8981(94)90263-1. PMID 7834862
- [Background] Lindblad A, Glaumann H, Strandvik B. Natural history of liver disease in cystic fibrosis. Hepatology. 1999 Nov;30(5):1151-8. doi: 10.1002/hep.510300527. PMID 10534335
- [Background] Colombo C, Battezzati PM. Hepatobiliary manifestations of cystic fibrosis. Eur J Gastroenterol Hepatol. 1996 Aug;8(8):748-54. PMID 8864670
- [Background] Sokol RJ, Durie PR. Recommendations for management of liver and biliary tract disease in cystic fibrosis. Cystic Fibrosis Foundation Hepatobiliary Disease Consensus Group. J Pediatr Gastroenterol Nutr. 1999;28 Suppl 1:S1-13. doi: 10.1097/00005176-199900001-00001. No abstract available. PMID 9934970
- [Background] Fishbein MH, Stevens WR. Rapid MRI using a modified Dixon technique: a non-invasive and effective method for detection and monitoring of fatty metamorphosis of the liver. Pediatr Radiol. 2001 Nov;31(11):806-9. doi: 10.1007/s002470100547. PMID 11692239
- [Background] Abdelmalek MF, Angulo P, Jorgensen RA, Sylvestre PB, Lindor KD. Betaine, a promising new agent for patients with nonalcoholic steatohepatitis: results of a pilot study. Am J Gastroenterol. 2001 Sep;96(9):2711-7. doi: 10.1111/j.1572-0241.2001.04129.x. PMID 11569700
- [Background] Moghaddami N, Costabile M, Grover PK, Jersmann HP, Huang ZH, Hii CS, Ferrante A. Unique effect of arachidonic acid on human neutrophil TNF receptor expression: up-regulation involving protein kinase C, extracellular signal-regulated kinase, and phospholipase A2. J Immunol. 2003 Sep 1;171(5):2616-24. doi: 10.4049/jimmunol.171.5.2616. PMID 12928414
- [Background] Miele L, Cordella-Miele E, Xing M, Frizzell R, Mukherjee AB. Cystic fibrosis gene mutation (deltaF508) is associated with an intrinsic abnormality in Ca2+-induced arachidonic acid release by epithelial cells. DNA Cell Biol. 1997 Jun;16(6):749-59. doi: 10.1089/dna.1997.16.749. PMID 9212168
- [Background] Levy E, Gurbindo C, Lacaille F, Paradis K, Thibault L, Seidman E. Circulating tumor necrosis factor-alpha levels and lipid abnormalities in patients with cystic fibrosis. Pediatr Res. 1993 Aug;34(2):162-6. doi: 10.1203/00006450-199308000-00011. PMID 8233719
- [Background] Rallidis LS, Paschos G, Liakos GK, Velissaridou AH, Anastasiadis G, Zampelas A. Dietary alpha-linolenic acid decreases C-reactive protein, serum amyloid A and interleukin-6 in dyslipidaemic patients. Atherosclerosis. 2003 Apr;167(2):237-42. doi: 10.1016/s0021-9150(02)00427-6. PMID 12818406
- [Background] De Vizia B, Raia V, Spano C, Pavlidis C, Coruzzo A, Alessio M. Effect of an 8-month treatment with omega-3 fatty acids (eicosapentaenoic and docosahexaenoic) in patients with cystic fibrosis. JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):52-7. doi: 10.1177/014860710302700152. PMID 12549599
- [Background] Kurlandsky LE, Bennink MR, Webb PM, Ulrich PJ, Baer LJ. The absorption and effect of dietary supplementation with omega-3 fatty acids on serum leukotriene B4 in patients with cystic fibrosis. Pediatr Pulmonol. 1994 Oct;18(4):211-7. doi: 10.1002/ppul.1950180404. PMID 7838619
- [Background] Tso P, Lam J, Simmonds WJ. The importance of the lysophosphatidylcholine and choline moiety of bile phosphatidylcholine in lymphatic transport of fat. Biochim Biophys Acta. 1978 Mar 30;528(3):364-72. doi: 10.1016/0005-2760(78)90025-5. PMID 638162
- [Background] Nilsson A, Borgstrom B. Absorption and metabolism of lecithin and lysolecithin by intestinal slices. Biochim Biophys Acta. 1967 Apr 4;137(2):240-54. doi: 10.1016/0005-2760(67)90100-2. No abstract available. PMID 6051560
- [Background] Nouri-Sorkhabi MH, Chapman BE, Kuchel PW, Gruca MA, Gaskin KJ. Parallel secretion of pancreatic phospholipase A(2), phospholipase A(1), lipase, and colipase in children with exocrine pancreatic dysfunction. Pediatr Res. 2000 Dec;48(6):735-40. doi: 10.1203/00006450-200012000-00006. PMID 11102539
- [Background] Lloyd-Still JD. Essential fatty acid deficiency and nutritional supplementation in cystic fibrosis. J Pediatr. 2002 Aug;141(2):157-9. doi: 10.1067/mpd.2002.126453. No abstract available. PMID 12183705
- [Background] Super M. Milestones in cystic fibrosis. Br Med Bull. 1992 Oct;48(4):717-37. doi: 10.1093/oxfordjournals.bmb.a072574. PMID 1281032
- [Background] Sheppard DN, Welsh MJ. Structure and function of the CFTR chloride channel. Physiol Rev. 1999 Jan;79(1 Suppl):S23-45. doi: 10.1152/physrev.1999.79.1.S23. PMID 9922375
- [Background] O'Riordan CR, Erickson A, Bear C, Li C, Manavalan P, Wang KX, Marshall J, Scheule RK, McPherson JM, Cheng SH, et al. Purification and characterization of recombinant cystic fibrosis transmembrane conductance regulator from Chinese hamster ovary and insect cells. J Biol Chem. 1995 Jul 14;270(28):17033-43. doi: 10.1074/jbc.270.28.17033. PMID 7542655
- [Background] Cobb BR, Ruiz F, King CM, Fortenberry J, Greer H, Kovacs T, Sorscher EJ, Clancy JP. A(2) adenosine receptors regulate CFTR through PKA and PLA(2). Am J Physiol Lung Cell Mol Physiol. 2002 Jan;282(1):L12-25. doi: 10.1152/ajplung.2002.282.1.L12. PMID 11741811
- [Background] Eidelman O, BarNoy S, Razin M, Zhang J, McPhie P, Lee G, Huang Z, Sorscher EJ, Pollard HB. Role for phospholipid interactions in the trafficking defect of Delta F508-CFTR. Biochemistry. 2002 Sep 17;41(37):11161-70. doi: 10.1021/bi020289s. PMID 12220181
- [Background] Weber AM, Roy CC, Chartrand L, Lepage G, Dufour OL, Morin CL, Lasalle R. Relationship between bile acid malabsorption and pancreatic insufficiency in cystic fibrosis. Gut. 1976 Apr;17(4):295-9. doi: 10.1136/gut.17.4.295. PMID 773791
- [Background] Goodchild MC, Murphy GM, Howell AM, Nutter SA, Anderson CM. Aspects of bile acid metabolism in cystic fibrosis. Arch Dis Child. 1975 Oct;50(10):769-78. doi: 10.1136/adc.50.10.769. PMID 1236566
- [Background] Roller RJ, Kern F. Minimal bile acid malabsorption and normal bile acid breath tests in cystic fibrosis and acquired pancreatic insufficiency. Gastroenterology. 1977 Apr;72(4 Pt 1):661-5. PMID 838220
- [Background] Harries JT, Muller DP, McCollum JP, Lipson A, Roma E, Norman AP. Intestinal bile salts in cystic fibrosis: studies in the patient and experimental animal. Arch Dis Child. 1979 Jan;54(1):19-24. doi: 10.1136/adc.54.1.19. PMID 420518
- [Background] van Berge Henegouwen GP, van der Werf SD, Ruben AT. Fatty acid composition of phospholipids in bile in man: promoting effect of deoxycholate on arachidonate. Clin Chim Acta. 1987 May 29;165(1):27-37. doi: 10.1016/0009-8981(87)90215-4. PMID 3111757
- [Background] Entenman C, Holloway RJ, Albright ML, Leong GF. Bile acids and lipid metabolism. II. Essential role of bile acids in bile phospholipid excretion. Arch Biochem Biophys. 1969 Mar;130(1):253-6. doi: 10.1016/0003-9861(69)90031-9. No abstract available. PMID 5778640
- [Background] Nilsson S, Schersten T. Importance of bile acids for phospholipid secretion into human hepatic bile. Gastroenterology. 1969 Nov;57(5):525-32. No abstract available. PMID 5348087
- [Background] Nilsson S, Schersten T. Influence of bile acids on the synthesis of biliary phospholipids in man. Eur J Clin Invest. 1970 Aug;1(2):109-11. doi: 10.1111/j.1365-2362.1970.tb00606.x. No abstract available. PMID 5450974
- [Background] Schersten T, Nilsson S, Cahlin E, Filipson M, Brodin-Persson G. Relationship between the biliary excretion of bile acids and the excretion of water, lecithin, and cholesterol in man. Eur J Clin Invest. 1971 Jan;1(4):242-7. doi: 10.1111/eci.1971.1.4.242. No abstract available. PMID 5549528
- [Background] Schersten T. Bile acids as a determining factor for synthesis and excretion of human bile lecithin. Helv Med Acta. 1973 Sep;37(2):161-8. No abstract available. PMID 4748925
- [Background] LeBlanc MJ, Gavino V, Perea A, Yousef IM, Levy E, Tuchweber B. The role of dietary choline in the beneficial effects of lecithin on the secretion of biliary lipids in rats. Biochim Biophys Acta. 1998 Aug 28;1393(2-3):223-34. doi: 10.1016/s0005-2760(98)00072-1. PMID 9748591
- [Background] Smit JJ, Schinkel AH, Oude Elferink RP, Groen AK, Wagenaar E, van Deemter L, Mol CA, Ottenhoff R, van der Lugt NM, van Roon MA, et al. Homozygous disruption of the murine mdr2 P-glycoprotein gene leads to a complete absence of phospholipid from bile and to liver disease. Cell. 1993 Nov 5;75(3):451-62. doi: 10.1016/0092-8674(93)90380-9. PMID 8106172
- [Background] Wibom R, Hultman E. ATP production rate in mitochondria isolated from microsamples of human muscle. Am J Physiol. 1990 Aug;259(2 Pt 1):E204-9. doi: 10.1152/ajpendo.1990.259.2.E204. PMID 2382713
- [Background] Blomstrand E, Ekblom B, Newsholme EA. Maximum activities of key glycolytic and oxidative enzymes in human muscle from differently trained individuals. J Physiol. 1986 Dec;381:111-8. doi: 10.1113/jphysiol.1986.sp016316. PMID 2957491
- [Background] Holloszy JO. Biochemical adaptations in muscle. Effects of exercise on mitochondrial oxygen uptake and respiratory enzyme activity in skeletal muscle. J Biol Chem. 1967 May 10;242(9):2278-82. No abstract available. PMID 4290225
- [Background] von Ruecker AA, Bertele R, Harms HK. Calcium metabolism and cystic fibrosis: mitochondrial abnormalities suggest a modification of the mitochondrial membrane. Pediatr Res. 1984 Jul;18(7):594-9. doi: 10.1203/00006450-198407000-00005. PMID 6206464
- [Background] Orenstein DM, Franklin BA, Doershuk CF, Hellerstein HK, Germann KJ, Horowitz JG, Stern RC. Exercise conditioning and cardiopulmonary fitness in cystic fibrosis. The effects of a three-month supervised running program. Chest. 1981 Oct;80(4):392-8. doi: 10.1378/chest.80.4.392. PMID 7023863
- [Background] Salh W, Bilton D, Dodd M, Webb AK. Effect of exercise and physiotherapy in aiding sputum expectoration in adults with cystic fibrosis. Thorax. 1989 Dec;44(12):1006-8. doi: 10.1136/thx.44.12.1006. PMID 2617441
- [Background] Nixon PA, Orenstein DM, Kelsey SF, Doershuk CF. The prognostic value of exercise testing in patients with cystic fibrosis. N Engl J Med. 1992 Dec 17;327(25):1785-8. doi: 10.1056/NEJM199212173272504. PMID 1435933
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Ward SA, Tomezsko JL, Holsclaw DS, Paolone AM. Energy expenditure and substrate utilization in adults with cystic fibrosis and diabetes mellitus. Am J Clin Nutr. 1999 May;69(5):913-9. doi: 10.1093/ajcn/69.5.913. PMID 10232630
- [Background] Buchdahl RM, Cox M, Fulleylove C, Marchant JL, Tomkins AM, Brueton MJ, Warner JO. Increased resting energy expenditure in cystic fibrosis. J Appl Physiol (1985). 1988 May;64(5):1810-6. doi: 10.1152/jappl.1988.64.5.1810. PMID 3391885
- [Background] Thomson MA, Wilmott RW, Wainwright C, Masters B, Francis PJ, Shepherd RW. Resting energy expenditure, pulmonary inflammation, and genotype in the early course of cystic fibrosis. J Pediatr. 1996 Sep;129(3):367-73. doi: 10.1016/s0022-3476(96)70068-9. PMID 8804325
- [Background] Fried MD, Durie PR, Tsui LC, Corey M, Levison H, Pencharz PB. The cystic fibrosis gene and resting energy expenditure. J Pediatr. 1991 Dec;119(6):913-6. doi: 10.1016/s0022-3476(05)83042-2. PMID 1960606
- [Background] Pencharz PB, Durie PR. Pathogenesis of malnutrition in cystic fibrosis, and its treatment. Clin Nutr. 2000 Dec;19(6):387-94. doi: 10.1054/clnu.1999.0079. PMID 11104588
- [Background] Bent ED, Bell JD. Quantification of the interactions among fatty acid, lysophosphatidylcholine, calcium, dimyristoylphosphatidylcholine vesicles, and phospholipase A2. Biochim Biophys Acta. 1995 Feb 9;1254(3):349-60. doi: 10.1016/0005-2760(94)00201-9. PMID 7857976
- [Background] Seid M, Varni JW, Segall D, Kurtin PS. Health-related quality of life as a predictor of pediatric healthcare costs: a two-year prospective cohort analysis. Health Qual Life Outcomes. 2004 Sep 10;2:48. doi: 10.1186/1477-7525-2-48. PMID 15361252
- [Background] Quittner AL. Measurement of quality of life in cystic fibrosis. Curr Opin Pulm Med. 1998 Nov;4(6):326-31. doi: 10.1097/00063198-199811000-00003. PMID 10813210
- [Background] Quittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of The Cystic Fibrosis Questionnaire in the United States: a health-related quality-of-life measure for cystic fibrosis. Chest. 2005 Oct;128(4):2347-54. doi: 10.1378/chest.128.4.2347. PMID 16236893
- [Background] Aris RM, Merkel PA, Bachrach LK, Borowitz DS, Boyle MP, Elkin SL, Guise TA, Hardin DS, Haworth CS, Holick MF, Joseph PM, O'Brien K, Tullis E, Watts NB, White TB. Guide to bone health and disease in cystic fibrosis. J Clin Endocrinol Metab. 2005 Mar;90(3):1888-96. doi: 10.1210/jc.2004-1629. Epub 2004 Dec 21. PMID 15613415
- [Background] Rovner AJ, Zemel BS, Leonard MB, Schall JI, Stallings VA. Mild to moderate cystic fibrosis is not associated with increased fracture risk in children and adolescents. J Pediatr. 2005 Sep;147(3):327-31. doi: 10.1016/j.jpeds.2005.04.015. PMID 16182670
- [Background] Baggio B. Fatty acids, calcium and bone metabolism. J Nephrol. 2002 Nov-Dec;15(6):601-4. PMID 12495271
- [Background] Watkins BA, Li Y, Seifert MF. Nutraceutical fatty acids as biochemical and molecular modulators of skeletal biology. J Am Coll Nutr. 2001 Oct;20(5 Suppl):410S-416S; discussion 417S-420S. doi: 10.1080/07315724.2001.10719177. PMID 11603651
- [Background] Albertazzi P, Coupland K. Polyunsaturated fatty acids. Is there a role in postmenopausal osteoporosis prevention? Maturitas. 2002 May 20;42(1):13-22. doi: 10.1016/s0378-5122(02)00022-1. PMID 12020975
- [Background] Kruger MC, Coetzer H, de Winter R, Gericke G, van Papendorp DH. Calcium, gamma-linolenic acid and eicosapentaenoic acid supplementation in senile osteoporosis. Aging (Milano). 1998 Oct;10(5):385-94. doi: 10.1007/BF03339885. PMID 9932142
- [Background] Bassey EJ, Littlewood JJ, Rothwell MC, Pye DW. Lack of effect of supplementation with essential fatty acids on bone mineral density in healthy pre- and postmenopausal women: two randomized controlled trials of Efacal v. calcium alone. Br J Nutr. 2000 Jun;83(6):629-35. doi: 10.1017/s0007114500000805. PMID 10911771
- [Background] Anthony H, Paxton S, Bines J, Phelan P. Psychosocial predictors of adherence to nutritional recommendations and growth outcomes in children with cystic fibrosis. J Psychosom Res. 1999 Dec;47(6):623-34. doi: 10.1016/s0022-3999(99)00065-3. PMID 10661608
- [Background] Lemanek KL, Kamps J, Chung NB. Empirically supported treatments in pediatric psychology: regimen adherence. J Pediatr Psychol. 2001 Jul-Aug;26(5):253-75. doi: 10.1093/jpepsy/26.5.253. PMID 11390568
- [Background] Weinstein AG, Cuskey W. Theophylline compliance in asthmatic children. Ann Allergy. 1985 Jan;54(1):19-24. PMID 3966686
- [Background] da Costa IG, Rapoff MA, Lemanek K, Goldstein GL. Improving adherence to medication regimens for children with asthma and its effect on clinical outcome. J Appl Behav Anal. 1997 Winter;30(4):687-91. doi: 10.1901/jaba.1997.30-687. PMID 9433792
- [Background] Wysocki T, Green L, Huxtable K. Blood glucose monitoring by diabetic adolescents: compliance and metabolic control. Health Psychol. 1989;8(3):267-84. doi: 10.1037//0278-6133.8.3.267. PMID 2767019
- [Background] Tucker CM, Petersen S, Herman KC, Fennell RS, Bowling B, Pedersen T, Vosmik JR. Self-regulation predictors of medication adherence among ethnically different pediatric patients with renal transplants. J Pediatr Psychol. 2001 Dec;26(8):455-64. doi: 10.1093/jpepsy/26.8.455. PMID 11700330
- [Background] Lemanek K. Adherence issues in the medical management of asthma. J Pediatr Psychol. 1990 Aug;15(4):437-58. doi: 10.1093/jpepsy/15.4.437. PMID 2258794
- [Background] Stark LJ, Bowen AM, Tyc VL, Evans S, Passero MA. A behavioral approach to increasing calorie consumption in children with cystic fibrosis. J Pediatr Psychol. 1990 Jun;15(3):309-26. doi: 10.1093/jpepsy/15.3.309. PMID 2380876
- [Background] Stark LJ, Knapp LG, Bowen AM, Powers SW, Jelalian E, Evans S, Passero MA, Mulvihill MM, Hovell M. Increasing calorie consumption in children with cystic fibrosis: replication with 2-year follow-up. J Appl Behav Anal. 1993 Winter;26(4):435-50. doi: 10.1901/jaba.1993.26-435. PMID 8307828
- [Background] Stark LJ, Mulvihill MM, Powers SW, Jelalian E, Keating K, Creveling S, Byrnes-Collins B, Harwood I, Passero MA, Light M, Miller DL, Hovell MF. Behavioral intervention to improve calorie intake of children with cystic fibrosis: treatment versus wait list control. J Pediatr Gastroenterol Nutr. 1996 Apr;22(3):240-53. doi: 10.1097/00005176-199604000-00005. PMID 8708877
- [Background] Stark LJ, Hommel KA, Mackner LM, Janicke DM, Davis AM, Pfefferkorn M, Crandall W, Heubi J. Randomized trial comparing two methods of increasing dietary calcium intake in children with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2005 Apr;40(4):501-7. doi: 10.1097/01.mpg.0000157913.32465.45. PMID 15795602
- [Background] Stark LJ, Janicke DM, McGrath AM, Mackner LM, Hommel KA, Lovell D. Prevention of osteoporosis: a randomized clinical trial to increase calcium intake in children with juvenile rheumatoid arthritis. J Pediatr Psychol. 2005 Jul-Aug;30(5):377-86. doi: 10.1093/jpepsy/jsi061. Epub 2005 Feb 23. PMID 15944165
- [Background] Borowitz D, Baker RD, Stallings V. Consensus report on nutrition for pediatric patients with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2002 Sep;35(3):246-59. doi: 10.1097/00005176-200209000-00004. No abstract available. PMID 12352509
- [Background] Tomezsko JL, Stallings VA, Scanlin TF. Dietary intake of healthy children with cystic fibrosis compared with normal control children. Pediatrics. 1992 Oct;90(4):547-53. PMID 1408508
- [Background] Zemel BS, Kawchak DA, Cnaan A, Zhao H, Scanlin TF, Stallings VA. Prospective evaluation of resting energy expenditure, nutritional status, pulmonary function, and genotype in children with cystic fibrosis. Pediatr Res. 1996 Oct;40(4):578-86. doi: 10.1203/00006450-199610000-00011. PMID 8888286
- [Background] Tomezsko JL, Stallings VA, Kawchak DA, Goin JE, Diamond G, Scanlin TF. Energy expenditure and genotype of children with cystic fibrosis. Pediatr Res. 1994 Apr;35(4 Pt 1):451-60. doi: 10.1203/00006450-199404000-00013. PMID 7519343
- [Background] Tomezsko JL, Scanlin TF, Stallings VA. Body composition of children with cystic fibrosis with mild clinical manifestations compared with normal children. Am J Clin Nutr. 1994 Jan;59(1):123-8. doi: 10.1093/ajcn/59.1.123. PMID 8279392
- [Background] Stettler N, Kawchak DA, Boyle LL, Propert KJ, Scanlin TF, Stallings VA, Zemel BS. Prospective evaluation of growth, nutritional status, and body composition in children with cystic fibrosis. Am J Clin Nutr. 2000 Aug;72(2):407-13. doi: 10.1093/ajcn/72.2.407. PMID 10919935
- [Background] Stallings VA, Fung EB, Hofley PM, Scanlin TF. Acute pulmonary exacerbation is not associated with increased energy expenditure in children with cystic fibrosis. J Pediatr. 1998 Mar;132(3 Pt 1):493-9. doi: 10.1016/s0022-3476(98)70026-5. PMID 9544907
- [Background] Stallings VA, Tomezsko JL, Schall JI, Mascarenhas MR, Stettler N, Scanlin TF, Zemel BS. Adolescent development and energy expenditure in females with cystic fibrosis. Clin Nutr. 2005 Oct;24(5):737-45. doi: 10.1016/j.clnu.2005.02.005. Epub 2005 Apr 8. PMID 16182037
- [Background] Fung EB, Barden EM, Wasserman D, Zemel BS, Heinrich BT, Scanlin TF, Stallings VA. A six-month study of growth and energy expenditure in children with cystic fibrosis taking a pulmonary inhalation medication (rhDNase). J Am Coll Nutr. 1999 Aug;18(4):330-8. doi: 10.1080/07315724.1999.10718872. PMID 12038476
- [Background] Zemel BS, Jawad AF, FitzSimmons S, Stallings VA. Longitudinal relationship among growth, nutritional status, and pulmonary function in children with cystic fibrosis: analysis of the Cystic Fibrosis Foundation National CF Patient Registry. J Pediatr. 2000 Sep;137(3):374-80. doi: 10.1067/mpd.2000.107891. PMID 10969263
- [Background] Cohen JR, Schall JI, Ittenbach RF, Zemel BS, Stallings VA. Fecal elastase: pancreatic status verification and influence on nutritional status in children with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2005 Apr;40(4):438-44. doi: 10.1097/01.mpg.0000158222.23181.1c. PMID 15795591
- [Background] Birch LL, Birch D, Marlin DW, Kramer L. Effects of instrumental consumption on children's food preference. Appetite. 1982 Jun;3(2):125-34. doi: 10.1016/s0195-6663(82)80005-6. No abstract available. PMID 7137991
- [Background] Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, Flegal KM, Guo SS, Wei R, Mei Z, Curtin LR, Roche AF, Johnson CL. CDC growth charts: United States. Adv Data. 2000 Jun 8;(314):1-27. PMID 11183293
- [Background] Koc H, Mar MH, Ranasinghe A, Swenberg JA, Zeisel SH. Quantitation of choline and its metabolites in tissues and foods by liquid chromatography/electrospray ionization-isotope dilution mass spectrometry. Anal Chem. 2002 Sep 15;74(18):4734-40. doi: 10.1021/ac025624x. PMID 12349977
- [Background] Han X, Gross RW. Electrospray ionization mass spectroscopic analysis of human erythrocyte plasma membrane phospholipids. Proc Natl Acad Sci U S A. 1994 Oct 25;91(22):10635-9. doi: 10.1073/pnas.91.22.10635. PMID 7938005
- [Background] Han X. Characterization and direct quantitation of ceramide molecular species from lipid extracts of biological samples by electrospray ionization tandem mass spectrometry. Anal Biochem. 2002 Mar 15;302(2):199-212. doi: 10.1006/abio.2001.5536. PMID 11878798
- [Background] Blom TS, Koivusalo M, Kuismanen E, Kostiainen R, Somerharju P, Ikonen E. Mass spectrometric analysis reveals an increase in plasma membrane polyunsaturated phospholipid species upon cellular cholesterol loading. Biochemistry. 2001 Dec 4;40(48):14635-44. doi: 10.1021/bi0156714. PMID 11724577
- [Background] Liebisch G, Drobnik W, Lieser B, Schmitz G. High-throughput quantification of lysophosphatidylcholine by electrospray ionization tandem mass spectrometry. Clin Chem. 2002 Dec;48(12):2217-24. PMID 12446479
- [Background] BLIGH EG, DYER WJ. A rapid method of total lipid extraction and purification. Can J Biochem Physiol. 1959 Aug;37(8):911-7. doi: 10.1139/o59-099. No abstract available. PMID 13671378
- [Background] Agren JJ, Julkunen A, Penttila I. Rapid separation of serum lipids for fatty acid analysis by a single aminopropyl column. J Lipid Res. 1992 Dec;33(12):1871-6. PMID 1479296
- [Background] Duffin K, Obukowicz M, Raz A, Shieh JJ. Electrospray/tandem mass spectrometry for quantitative analysis of lipid remodeling in essential fatty acid deficient mice. Anal Biochem. 2000 Mar 15;279(2):179-88. doi: 10.1006/abio.1999.4452. PMID 10706787
- [Background] Brugger B, Erben G, Sandhoff R, Wieland FT, Lehmann WD. Quantitative analysis of biological membrane lipids at the low picomole level by nano-electrospray ionization tandem mass spectrometry. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2339-44. doi: 10.1073/pnas.94.6.2339. PMID 9122196
- [Background] Koivusalo M, Haimi P, Heikinheimo L, Kostiainen R, Somerharju P. Quantitative determination of phospholipid compositions by ESI-MS: effects of acyl chain length, unsaturation, and lipid concentration on instrument response. J Lipid Res. 2001 Apr;42(4):663-72. PMID 11290839
- [Background] DeLong CJ, Baker PR, Samuel M, Cui Z, Thomas MJ. Molecular species composition of rat liver phospholipids by ESI-MS/MS: the effect of chromatography. J Lipid Res. 2001 Dec;42(12):1959-68. PMID 11734568
- [Background] Hollis BW, Kamerud JQ, Selvaag SR, Lorenz JD, Napoli JL. Determination of vitamin D status by radioimmunoassay with an 125I-labeled tracer. Clin Chem. 1993 Mar;39(3):529-33. PMID 8448871
- [Background] Hollis BW, Kamerud JQ, Kurkowski A, Beaulieu J, Napoli JL. Quantification of circulating 1,25-dihydroxyvitamin D by radioimmunoassay with 125I-labeled tracer. Clin Chem. 1996 Apr;42(4):586-92. PMID 8605676
- [Background] Hauschka PV, Lian JB, Cole DE, Gundberg CM. Osteocalcin and matrix Gla protein: vitamin K-dependent proteins in bone. Physiol Rev. 1989 Jul;69(3):990-1047. doi: 10.1152/physrev.1989.69.3.990. No abstract available. PMID 2664828
- [Background] Gallop PM, Lian JB, Hauschka PV. Carboxylated calcium-binding proteins and vitamin K. N Engl J Med. 1980 Jun 26;302(26):1460-6. doi: 10.1056/NEJM198006263022608. No abstract available. PMID 6990261
- [Background] Bikle DD. Biochemical markers in the assessment of bone disease. Am J Med. 1997 Nov;103(5):427-36. doi: 10.1016/s0002-9343(97)00137-x. PMID 9375712
- [Background] Price CP. Multiple forms of human serum alkaline phosphatase: detection and quantitation. Ann Clin Biochem. 1993 Jul;30 ( Pt 4):355-72. doi: 10.1177/000456329303000403. No abstract available. PMID 8379650
- [Background] ATS statement--Snowbird workshop on standardization of spirometry. Am Rev Respir Dis. 1979 May;119(5):831-8. doi: 10.1164/arrd.1979.119.5.831. No abstract available. PMID 453705
- [Background] Weir JB. New methods for calculating metabolic rate with special reference to protein metabolism. 1949. Nutrition. 1990 May-Jun;6(3):213-21. No abstract available. PMID 2136000
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Background] Feskanich D, Buzzard IM, Welch BT, Asp EH, Dieleman LS, Chong KR, Bartsch GE. Comparison of a computerized and a manual method of food coding for nutrient intake studies. J Am Diet Assoc. 1988 Oct;88(10):1263-7. PMID 3171019
- [Background] Himes JH, Roche AF, Thissen D, Moore WM. Parent-specific adjustments for evaluation of recumbent length and stature of children. Pediatrics. 1985 Feb;75(2):304-13. PMID 3969331
- [Background] Brook CG. Determination of body composition of children from skinfold measurements. Arch Dis Child. 1971 Apr;46(246):182-4. doi: 10.1136/adc.46.246.182. PMID 5576028
- [Background] Slaughter MH, Lohman TG, Boileau RA, Horswill CA, Stillman RJ, Van Loan MD, Bemben DA. Skinfold equations for estimation of body fatness in children and youth. Hum Biol. 1988 Oct;60(5):709-23. No abstract available. PMID 3224965
- [Background] Wahner HW, Looker A, Dunn WL, Walters LC, Hauser MF, Novak C. Quality control of bone densitometry in a national health survey (NHANES III) using three mobile examination centers. J Bone Miner Res. 1994 Jun;9(6):951-60. doi: 10.1002/jbmr.5650090621. PMID 8079669
- [Background] Faulkner KG, Gluer CC, Grampp S, Genant HK. Cross-calibration of liquid and solid QCT calibration standards: corrections to the UCSF normative data. Osteoporos Int. 1993 Jan;3(1):36-42. doi: 10.1007/BF01623175. PMID 8422515
- [Background] Louis O, Soykens S, Willnecker J, Van den Winkel P, Osteaux M. Cortical and total bone mineral content of the radius: accuracy of peripheral computed tomography. Bone. 1996 May;18(5):467-72. doi: 10.1016/8756-3282(96)00040-3. PMID 8739905
- [Background] Braun MJ, Meta MD, Schneider P, Reiners C. Clinical evaluation of a high-resolution new peripheral quantitative computerized tomography (pQCT) scanner for the bone densitometry at the lower limbs. Phys Med Biol. 1998 Aug;43(8):2279-94. doi: 10.1088/0031-9155/43/8/020. PMID 9725604
- [Background] Henderson RC, Lin PP, Greene WB. Bone-mineral density in children and adolescents who have spastic cerebral palsy. J Bone Joint Surg Am. 1995 Nov;77(11):1671-81. doi: 10.2106/00004623-199511000-00005. PMID 7593076
- [Background] Lappe JM, Stegman M, Davies KM, Barber S, Recker RR. A prospective study of quantitative ultrasound in children and adolescents. J Clin Densitom. 2000 Summer;3(2):167-75. doi: 10.1385/jcd:3:2:167. PMID 10873227
- [Background] Lum CK, Wang MC, Moore E, Wilson DM, Marcus R, Bachrach LK. A comparison of calcaneus ultrasound and dual X-ray absorptiometry in healthy North American youths and young adults. J Clin Densitom. 1999 Winter;2(4):403-11. doi: 10.1016/s1094-6950(06)60406-x. PMID 10677794
- [Background] Falcini F, Bindi G, Ermini M, Galluzzi F, Poggi G, Rossi S, Masi L, Cimaz R, Brandi ML. Comparison of quantitative calcaneal ultrasound and dual energy X-ray absorptiometry in the evaluation of osteoporotic risk in children with chronic rheumatic diseases. Calcif Tissue Int. 2000 Jul;67(1):19-23. doi: 10.1007/s00223001090. PMID 10908407
- [Background] Resch H, Newrkla S, Grampp S, Resch A, Zapf S, Piringer S, Hockl A, Weiss P. Ultrasound and X-ray-based bone densitometry in patients with anorexia nervosa. Calcif Tissue Int. 2000 May;66(5):338-41. doi: 10.1007/s002230010070. PMID 10773102
- [Background] Grampp S, Henk CB, Fuerst TP, Lu Y, Bader TR, Kainberger F, Genant HK, Imhof H. Diagnostic agreement of quantitative sonography of the calcaneus with dual X-ray absorptiometry of the spine and femur. AJR Am J Roentgenol. 1999 Aug;173(2):329-34. doi: 10.2214/ajr.173.2.10430129.
- [Background] Gnudi S, Ripamonti C, Malavolta N. Quantitative ultrasound and bone densitometry to evaluate the risk of nonspine fractures: a prospective study. Osteoporos Int. 2000;11(6):518-23. doi: 10.1007/s001980070095. PMID 10982168
- [Background] Mughal MZ, Langton CM, Utretch G, Morrison J, Specker BL. Comparison between broad-band ultrasound attenuation of the calcaneum and total body bone mineral density in children. Acta Paediatr. 1996 Jun;85(6):663-5. doi: 10.1111/j.1651-2227.1996.tb14119.x. PMID 8816199
- [Background] Leggin BG, Neuman RM, Iannotti JP, Williams GR, Thompson EC. Intrarater and interrater reliability of three isometric dynamometers in assessing shoulder strength. J Shoulder Elbow Surg. 1996 Jan-Feb;5(1):18-24. doi: 10.1016/s1058-2746(96)80026-7. PMID 8919438
- [Background] Vandenborne K, Elliott MA, Walter GA, Abdus S, Okereke E, Shaffer M, Tahernia D, Esterhai JL. Longitudinal study of skeletal muscle adaptations during immobilization and rehabilitation. Muscle Nerve. 1998 Aug;21(8):1006-12. doi: 10.1002/(sici)1097-4598(199808)21:83.0.co;2-c. PMID 9655118
- [Background] Schall JI, Semeao EJ, Stallings VA, Zemel BS. Self-assessment of sexual maturity status in children with Crohn's disease. J Pediatr. 2002 Aug;141(2):223-9. doi: 10.1067/mpd.2002.125907. PMID 12183718
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Modi AC, Quittner AL. Validation of a disease-specific measure of health-related quality of life for children with cystic fibrosis. J Pediatr Psychol. 2003 Dec;28(8):535-45. doi: 10.1093/jpepsy/jsg044. PMID 14602844
- [Background] Zhang J, Quan H, Ng J, Stepanavage ME. Some statistical methods for multiple endpoints in clinical trials. Control Clin Trials. 1997 Jun;18(3):204-21. doi: 10.1016/s0197-2456(96)00129-8. PMID 9204221
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Derived] Tindall A, Mascarenhas M, Maqbool A, Stallings VA. Lysophosphatidylcholine-Rich Nutrition Therapy Increased Gut Absorption of Coingested Dietary Fat: a Randomized Controlled Trial. Curr Dev Nutr. 2023 Jul 31;7(9):101985. doi: 10.1016/j.cdnut.2023.101985. eCollection 2023 Sep. PMID 37671264
- [Derived] Stallings VA, Tindall AM, Mascarenhas MR, Maqbool A, Schall JI. Improved residual fat malabsorption and growth in children with cystic fibrosis treated with a novel oral structured lipid supplement: A randomized controlled trial. PLoS One. 2020 May 8;15(5):e0232685. doi: 10.1371/journal.pone.0232685. eCollection 2020. PMID 32384122
- [Derived] Stallings VA, Schall JI, Maqbool A, Mascarenhas MR, Alshaikh BN, Dougherty KA, Hommel K, Ryan J, Elci OU, Shaw WA. Effect of Oral Lipid Matrix Supplement on Fat Absorption in Cystic Fibrosis: A Randomized Placebo-Controlled Trial. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):676-680. doi: 10.1097/MPG.0000000000001213. PMID 27050056
- [Derived] Schall JI, Mascarenhas MR, Maqbool A, Dougherty KA, Elci O, Wang DJ, Altes TA, Hommel KA, Shaw W, Moore J, Stallings VA. Choline Supplementation With a Structured Lipid in Children With Cystic Fibrosis: A Randomized Placebo-Controlled Trial. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):618-26. doi: 10.1097/MPG.0000000000001004. PMID 26465792
- [Derived] Groleau V, Schall JI, Dougherty KA, Latham NE, Maqbool A, Mascarenhas MR, Stallings VA. Effect of a dietary intervention on growth and energy expenditure in children with cystic fibrosis. J Cyst Fibros. 2014 Sep;13(5):572-8. doi: 10.1016/j.jcf.2014.01.009. Epub 2014 Feb 8. PMID 24518280
- [Derived] Bertolaso C, Groleau V, Schall JI, Maqbool A, Mascarenhas M, Latham NE, Dougherty KA, Stallings VA. Fat-soluble vitamins in cystic fibrosis and pancreatic insufficiency: efficacy of a nutrition intervention. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):443-8. doi: 10.1097/MPG.0000000000000272. PMID 24345827